CLINICAL TRIAL: NCT00282347
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Rituximab in Subjects With ISN/RPS Class III or IV Lupus Nephritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Rituximab in Subjects With International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 Class III or IV Lupus Nephritis
Acronym: LUNAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U2970g
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Lupus Nephritis
Keywords: Class IV LN; Lupus; LUNAR; LN
MeSH Terms: conditions — Lupus Nephritis | interventions — Rituximab; Mycophenolic Acid; Methylprednisolone; Diphenhydramine; Acetaminophen; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Experimental): Participants received rituximab 1000 mg intravenously (IV) on Days 1, 15, 168, and 182. They also received mycophenolate mofetil, methylprednisolone, diphenhydramine, acetaminophen, and prednisone; see the Detailed Description for details.
  Interventions: Drug: Rituximab; Drug: Mycophenolate mofetil; Drug: Methylprednisolone; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Prednisone
- Placebo (Placebo Comparator): Participants received placebo intravenously (IV) on Days 1, 15, 168, and 182. They also received mycophenolate mofetil, methylprednisolone, diphenhydramine, acetaminophen, and prednisone; see the Detailed Description for details.
  Interventions: Drug: Placebo; Drug: Mycophenolate mofetil; Drug: Methylprednisolone; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Rituximab was provided as a sterile solution for injection.
  Other Names: Rituxan; MabThera; Zytux
  Arms: Rituximab
Drug: Placebo — Placebo was provided as a sterile solution for injection.
  Arms: Placebo
Drug: Mycophenolate mofetil
  Other Names: CellCept
Drug: Methylprednisolone
Drug: Diphenhydramine
Drug: Acetaminophen
Drug: Prednisone

SUMMARY:
This was a Phase III, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of rituximab in combination with mycophenolate mofetil (MMF) compared with placebo in combination with MMF in subjects diagnosed with International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 Class III or IV lupus nephritis.

DETAILED DESCRIPTION:
In addition to receiving study drug (rituximab or placebo), participants in each treatment group received mycophenolate mofetil at a starting dose of 1500 mg/day IV in 3 divided doses and were titrated up by 500 mg/week to 3000 mg/day by Week 4, as tolerated. Participants in each treatment group also received methylprednisolone 1000 mg IV prior to and 3 days following the first study drug infusion and methylprednisolone 100 mg IV prior to the other study drug infusions. Participants in each treatment group also received diphenhydramine 50 mg orally and acetaminophen 1000 mg orally 30-60 minutes prior to each study drug infusion. From Days 2 to 16, participants in each treatment group received prednisone 0.75 mg/kg/day orally (maximum dose of 60 mg) except on the day of the second methylprednisolone dose. On Day 16, a taper was initiated to achieve a dose of 10 mg/day by Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE) according to current American College of Rheumatology (ACR) criteria.
* Diagnosis of International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 Class III or IV lupus nephritis (LN), with either active or active/chronic disease.
* Proteinuria.
* 16-75 years of age.

Exclusion Criteria:

* Retinitis, poorly controlled seizure disorder, acute confusional state, myelitis, stroke or stroke syndrome, cerebellar ataxia, or dementia that is currently active and resulting from SLE.
* Unstable subjects with thrombocytopenia experiencing or at high risk for developing clinically significant bleeding or organ dysfunction requiring therapies such as plasmapheresis or acute blood or platelet transfusions.
* Lack of peripheral venous access.
* Pregnancy or lactation.
* History of severe allergic or anaphylactic reactions to monoclonal antibodies.
* Significant or uncontrolled medical disease in any organ system not related to SLE or LN, which, in the investigator's opinion, would preclude subject participation.
* Concomitant chronic conditions, excluding SLE (eg, asthma, Crohn's disease) that require oral or systemic corticosteroid use in the 52 weeks prior to screening.
* History of renal transplant.
* Known human immunodeficiency virus (HIV) infection.
* Known active infection of any kind (but excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with intravenous anti-infectives within 4 weeks of randomization or oral anti-infectives within 2 weeks of randomization.
* History of deep space infection within 1 year of screening.
* History of serious recurrent or chronic infection.
* History of cancer, including solid tumors, hematological malignancies, and carcinoma in situ (except basal cell carcinomas of the skin that have been treated or excised and have resolved).
* Currently active alcohol or drug abuse or history of alcohol or drug abuse within 52 weeks prior to screening.
* Major surgery requiring hospitalization within 4 weeks of screening (excluding diagnostic surgery).
* Treatment with cyclophosphamide or calcineurin inhibitors within the 90 days prior to screening.
* Use of mycophenolate mofetil (MMF) at a dose of > 2 grams daily for longer than the 90 days prior to screening.
* Intolerance or history of allergic reaction to MMF.
* Intolerance or history of allergic reaction to both angiotensin-converting enzyme (ACE) inhibitors and angiotensin-receptor blockers.
* Use of oral prednisone (or corticosteroid equivalent) at a dose of > 20 mg/day for longer than the 14 days prior to screening.
* Previous treatment with CAMPATH-1H (alemtuzumab).
* Previous treatment with a B-cell targeted therapy.
* Treatment with any investigational agent (including biologic agents approved for other indications) within 28 days of the start of the screening period or 5 half-lives of the investigational drug (whichever is longer).
* Receipt of a live vaccine within the 28 days prior to screening.
* Intolerance or contraindication to oral or IV corticosteroids.
* Current therapy with a nonsteroidal anti-inflammatory agent.
* Positive hepatitis B sAg or hepatitis C serology.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brunetta, MD, Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Gomez Mendez LM, Cascino MD, Garg J, Katsumoto TR, Brakeman P, Dall'Era M, Looney RJ, Rovin B, Dragone L, Brunetta P. Peripheral Blood B Cell Depletion after Rituximab and Complete Response in Lupus Nephritis. Clin J Am Soc Nephrol. 2018 Oct 8;13(10):1502-1509. doi: 10.2215/CJN.01070118. Epub 2018 Aug 8. PMID 30089664
- [Derived] Wolf BJ, Spainhour JC, Arthur JM, Janech MG, Petri M, Oates JC. Development of Biomarker Models to Predict Outcomes in Lupus Nephritis. Arthritis Rheumatol. 2016 Aug;68(8):1955-63. doi: 10.1002/art.39623. PMID 26867033
- [Derived] Rovin BH, Furie R, Latinis K, Looney RJ, Fervenza FC, Sanchez-Guerrero J, Maciuca R, Zhang D, Garg JP, Brunetta P, Appel G; LUNAR Investigator Group. Efficacy and safety of rituximab in patients with active proliferative lupus nephritis: the Lupus Nephritis Assessment with Rituximab study. Arthritis Rheum. 2012 Apr;64(4):1215-26. doi: 10.1002/art.34359. Epub 2012 Jan 9. PMID 22231479

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Rituximab | Placebo
Started | 72 | 72
Completed | 67 | 63
Not Completed | 5 | 9
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 0 | 1
Period: Safety Follow-up Period
Arm/Group | Rituximab | Placebo
Started | 67 | 63
Completed | 64 | 57
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Deviation | 0 | 2
Period: B Cell Follow-up Period
Arm/Group | Rituximab | Placebo
Started | 20 | 4
Completed | 15 | 4
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Reason Not Specified | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Customized [Number; unit: participants]
  < 18 years | 2 | 1 | 3
  18 to < 35 years | 48 | 48 | 96
  35 to < 50 years | 18 | 19 | 37
  ≥ 50 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (9.6) | 29.4 (9.3) | 30.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 67 | 130
  Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Complete Renal Response (CRR), a Partial Renal Response (PRR), or no Renal Response (NRR) at Week 52
Description: A participant had a CRR if they met the following 3 criteria: (1) Normalization of serum creatinine (SC) as evidenced by a SC level ≤ the upper limit of the normal range of central laboratory values or a SC level ≤ 15% greater than Baseline, if Baseline SC was within the normal range of the central laboratory values; (2) Inactive urinary sediment (as evidenced by < 5 red blood cells/high-power field (RBCs/HPF) and absence of red cell casts; (3) Urinary protein (UP) to creatinine ratio (CR) < 0.5. A participant had a PRR if they met the following 3 criteria: (1) A SC level ≤ 15% above Baseline; (2) RBCs/HPF ≤ 50% above Baseline and no RBC casts; (3) 50% improvement in the UP to CR, with 1 of the following conditions met: If the Baseline UP to CR was ≤ 3.0, then a UP to CR of < 1.0 or if the Baseline UP to CR was > 3.0, then a UP to CR of ≤ 3.0. A participant had a NRR if they did not achieve either a CRR or PRR.
Time Frame: Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
Percentage of participants
  CRR | 26.4 | 30.6
  PRR | 30.6 | 15.3
  NRR | 43.1 | 54.2
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority or Other; p = 0.5538, Stratified Wilcoxon-Rank Sum Test

2. Secondary Outcome: Percentage of Participants Who Achieved a Complete Renal Response at Week 24 and Maintained it to Week 52
Description: A participant had a complete renal response if they met the following 3 criteria: (1) Normalization of serum creatinine as evidenced by a serum creatinine level ≤ the upper limit of the normal range of central laboratory values or a serum creatinine level ≤ 15% greater than Baseline, if Baseline serum creatinine was within the normal range of the central laboratory values; (2) Inactive urinary sediment (as evidenced by < 5 red blood cells/high-power field and absence of red cell casts; (3) Urinary protein to creatinine ratio < 0.5.
Time Frame: Week 24 to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
Percentage of participants | 1.4 | 6.9

3. Secondary Outcome: Percentage of Participants Who Achieved a Complete Renal Response at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
Percentage of participants | 26.4 | 30.6

4. Secondary Outcome: Percentage of Participants With a Baseline Urine Protein to Creatinine Ratio of > 3.0 Who Achieved a Urine Protein to Creatinine Ratio of < 1.0 at Week 52
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo). Only those participants with a Baseline urine protein to creatinine ratio of > 3.0 were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 38 | 41
Percentage of participants | 47.4 | 53.7

5. Secondary Outcome: British Isles Lupus Assessment Group (BILAG) Index Score Over 52 Weeks
Description: The BILAG Index assesses 86 clinical signs and symptoms and laboratory measures of systemic lupus erythematosus in 8 organ system domains: General, mucocutaneous, neurological, musculoskeletal, cardiorespiratory, vasculitis, renal, and hematologic. Most of the 86 items are rated on the following scale: 0=Not present, 1=Improving, 2=Same, 3=Worse, 4=New. Some items are rated as either Yes or No. A single alphabetic score of A (very active) through E (not or never active) for each of the 8 domains is determined from the rating of the individual items in each domain. The total BILAG score is the sum of the scores of the 8 domains where A=9, B=3, C=1, D=0, and E=0. The total score ranges from 0 to 72 with a higher score indicating greater lupus activity. To calculate a BILAG score over the 52 week treatment period of the study, the area under the response-time curve of BILAG scores assessed every 4 weeks was divided by the number of days in the time curve minus the Baseline BILAG score.
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
Units on a scale | -8.49 (5.79) | -8.58 (5.14)

6. Secondary Outcome: Time to Achieve a Complete Renal Response
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
Weeks | 11.99 [8.31 to NA] — The upper limit of the confidence interval could not be estimated due to too few events. | 12.12 [9.26 to 13.47]

7. Secondary Outcome: Change From Baseline in the Systemic Lupus Erythematosus Expanded Health Survey Physical Function Score at Week 52
Description: The systemic lupus erythematosus Expanded Health Survey is based on the Short Form 36 Health survey with additional questions specific to lupus. The physical function component score of the survey can range from 0-100. A higher score indicates better health. A positive change score indicates improvement.
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
Units on a scale | 4.8 (10.4) | 5.7 (9.4)

8. Secondary Outcome: Change From Baseline in Anti-double-stranded DNA at Week 52
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
IU/mL | 0.45 (0.35) | 1.06 (2.19)

9. Secondary Outcome: Change From Baseline in C3 and C4 Complement Levels at Week 52
Time Frame: Baseline to Week 52
Population: Intent-to-treat population: All randomized participants who received any amount of study drug (rituximab or placebo).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 72 | 72
mg/dL
  C3 Complement | 37.5 (28.7) | 25.9 (32.5)
  C4 Complement | 9.9 (7.5) | 6.6 (8.9)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (up to 7 years)
Description: Safety analysis population: All randomized subjects who receive any amount of study drug (rituximab or placebo).
  Adverse events reported for the B cell follow-up period only include adverse events that occurred in participants who were followed after the last participant reached study Week 78.
Groups:
- Rituximab - Treatment and Safety Follow-up Periods; Rituximab - B Cell Follow-up Period: Participants received rituximab 1000 mg intravenously (IV) on Days 1, 15, 168, and 182. They also received mycophenolate mofetil, methylprednisolone, diphenhydramine, acetaminophen, and prednisone; see the Detailed Description for details.
- Placebo - Treatment and Safety Follow-up Periods; Placebo - B Cell Follow-up Period: Participants received placebo intravenously (IV) on Days 1, 15, 168, and 182. They also received mycophenolate mofetil, methylprednisolone, diphenhydramine, acetaminophen, and prednisone; see the Detailed Description for details.
Arm/Group | Rituximab - Treatment and Safety Follow-up Periods | Placebo - Treatment and Safety Follow-up Periods | Rituximab - B Cell Follow-up Period | Placebo - B Cell Follow-up Period
Serious Adverse Events (participants affected / at risk) | 24/73 | 29/71 | 3/20 | 0/4
Other Adverse Events (participants affected / at risk) | 69/73 | 66/71 | 8/20 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab - Treatment and Safety Follow-up Periods (N=73) | Placebo - Treatment and Safety Follow-up Periods (N=71) | Rituximab - B Cell Follow-up Period (N=20) | Placebo - B Cell Follow-up Period (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 2 | 0 | 0
Drug Intolerance (General disorders) | 1 | 0 | 0 | 0
Generalized Oedema (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Antiphospholipid Syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial Infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Catheter Related Infection (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0
Genital Herpes (Infections and infestations) | 0 | 1 | 0 | 0
Histoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia Cryptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia Cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0 | 0
International Normalized Ratio Decreased (Investigations) | 0 | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 2 | 0 | 0
Vasculitis Cerebral (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypersensitive Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 3 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Malignant Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0
Vena Cava Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Pyelonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Nephrogenic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Renal transplant (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab - Treatment and Safety Follow-up Periods (N=73) | Placebo - Treatment and Safety Follow-up Periods (N=71) | Rituximab - B Cell Follow-up Period (N=20) | Placebo - B Cell Follow-up Period (N=4)
Anaemia (Blood and lymphatic system disorders) | 10 | 9 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 6 | 5 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 4 | 0 | 0
Cushingoid (Endocrine disorders) | 4 | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 3 | 4 | 0 | 0
Vision Blurred (Eye disorders) | 3 | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 28 | 28 | 0 | 0
Nausea (Gastrointestinal disorders) | 20 | 21 | 0 | 0
Vomiting (Gastrointestinal disorders) | 19 | 14 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 9 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 7 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 4 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 4 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 4 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Oedema Peripheral (General disorders) | 6 | 11 | 0 | 0
Oedema (General disorders) | 8 | 7 | 0 | 0
Chest Pain (General disorders) | 4 | 10 | 0 | 0
Pyrexia (General disorders) | 9 | 4 | 0 | 0
Chills (General disorders) | 2 | 4 | 0 | 0
Pain (General disorders) | 2 | 4 | 0 | 0
Seasonal Allergy (Immune system disorders) | 5 | 0 | 0 | 0
Fatigue (General disorders) | 12 | 9 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 23 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 17 | 20 | 3 | 0
Herpes Zoster (Infections and infestations) | 11 | 8 | 0 | 0
Gastroenteritis (Infections and infestations) | 8 | 7 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 5 | 1 | 0
Sinusitis (Infections and infestations) | 9 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 4 | 0 | 0
Oral Candidiasis (Infections and infestations) | 6 | 4 | 0 | 0
Candidiasis (Infections and infestations) | 4 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 4 | 0 | 0
Influenza (Infections and infestations) | 3 | 4 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 4 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 1 | 0 | 0
Blood Potassium Decreased (Investigations) | 1 | 4 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 10 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 3 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 17 | 18 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 16 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 9 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 11 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0
Headache (Nervous system disorders) | 26 | 19 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 5 | 0 | 0
Tremor (Nervous system disorders) | 3 | 5 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 5 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 5 | 0 | 0
Insomnia (Psychiatric disorders) | 10 | 14 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 8 | 0 | 0
Depression (Psychiatric disorders) | 5 | 6 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 13 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 6 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 8 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 8 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0
Hypertension (Vascular disorders) | 7 | 7 | 0 | 0
Hypotension (Vascular disorders) | 8 | 3 | 0 | 0
Pyelonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Ear infection (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Amenorrhoea (Endocrine disorders) | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.